CLINICAL TRIAL: NCT04567355
Title: Migraine Manager: An Individualized Self-Management Tool for Adolescents With Migraine (R01)
Brief Title: Migraine Manager (R01)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MM R01; R01NR019426 (NIH)
Record Dates: First submitted 2020-09-23; First posted 2020-09-28 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Migraine; Migraine Disorders
Keywords: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The study PI, statistician, co-investigators, and all personnel who are involved in endpoint assessments will be blinded. Only one team member (lead CRC) will have access to the assignment of each participant.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Migraine Manager (Experimental): The Migraine Manager portal intervention is comprised of 16 modules that are assigned in an individually tailored manner to participants based on their answers to a brief assessment battery. Once assessments are completed, a treatment plan consisting of recommended modules is automatically generated for patient and parent guidance, and the user is directed to the list of recommended modules. Participants will also complete online daily diaries for eight weeks.
  Interventions: Behavioral: Migraine Manager
- Attention Control (No Intervention): Participants in this arm will complete the online daily diaries for eight weeks (i.e., equal time as the Migraine Manager arm) through the portal but will be restricted from receiving intervention content; they will also receive equal number of communications via the portal as the Migraine Manager arm. Data from migraine daily diaries will not be available to AC participants or their clinicians as this would likely be used clinically and lead to contamination of the control arm resulting from varying levels of intervention across participants based on their data.

INTERVENTIONS:
Behavioral: Migraine Manager — Answers provided during the online assessment will result in certain intervention recommendations. Once assessments are completed, a treatment plan will be automatically generated for patient and parent guidance.
  Arms: Migraine Manager

SUMMARY:
The objective of this trial is to test whether an online tailored intervention, Migraine Manager, is efficacious in improving headache outcomes compared to an attention control intervention in adolescents with migraines. We will conduct a randomized clinical trial to compare a sample of 80 youth (ages 11 to 17) with migraine receiving the online tailored adherence intervention to 80 youth in an attention control group. We will test whether adherence to healthy habit (hydration, regular meals, exercise, sleep) recommendations serves as a mechanism for improved headache outcomes. Clinically meaningful outcomes will be assessed by reliable, valid, and sensitive measures. The primary outcome (i.e., number of headache days) will be assessed via online daily diary pre- and post-intervention, with additional follow-up at 3, 6, 9, and 12 months. Secondary outcomes include health-related quality of life and migraine disability.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of migraine using current International Classification of Headache Disorders Criteria (ICHD-3) for migraine with or without aura
* Frequency of 8 or more headaches per month
* Access to the internet whether public (e.g., library) or private (e.g., home, personal)
* English fluency for patient and caregiver

Exclusion Criteria:

* Patients with a diagnosis of pervasive developmental disorder as determined by medical chart review
* Patients with a diagnosis of or serious mental illness (e.g., psychotic disorder) as determined by medical chart review

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Headache frequency | 15 months
  Change in number of days with a headache

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Hommel, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Scott Powers, PhD, Study Chair — Children's Hospital Medical Center, Cincinnati; Andrew Hershey, MD, PhD, Study Chair — Children's Hospital Medical Center, Cincinnati; Susan LeCates, MSN, FNP, Study Chair — Children's Hospital Medical Center, Cincinnati; Marielle Kabbouche-Samaha, MD, Study Chair — Children's Hospital Medical Center, Cincinnati; James Peugh, PhD, Study Chair — Children's Hospital Medical Center, Cincinnati; Lee Ritterband, MD, Study Chair — University of Virginia
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No